CLINICAL TRIAL: NCT02150096
Title: Laser and and Ultrasound Effect on Pain and Disability in Women With Chronic Non-specific Low Back Pain: a Randomized Controlled Trial
Brief Title: Laser and Therapeutic Ultrasound in the Management of the Chronic Non-specific Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Ana Paula Fernandes A. Rubira, Doctor, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEP 390/10
Record Dates: First submitted 2014-03-07; First posted 2014-05-29 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Chronic Low Back Pain
Keywords: chronic non-specific low back pain; clinical trial; disability; women

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Continuous ultrasound group (Active Comparator): the group will be treated with 1,5 W/cm² 6 minutes in each side of the lumbar spine in 6 points around the lumbar spine
  Interventions: Other: pulsed ultrasound group; Other: low level laser therapy group
- Pulsed ultrasound group (Active Comparator): the group will be treated with 1,5 W/cm² 6 minutes in each side of the lumbar spine in 6 points around the lumbar spine
  Interventions: Other: continuous ultrasound group; Other: low level laser therapy group
- low level laser therapy group (Active Comparator): the group will be treated with 3J during 6 minutes in each side of the lumbar spine in 6 points around the lumbar spine
  Interventions: Other: continuous ultrasound group; Other: pulsed ultrasound group
- control group (No Intervention): group of women no treated, only evaluated in two moments and this group will be compared with orthers: laser, pulsed ultrasound and continuous ultrasound.

INTERVENTIONS:
Other: continuous ultrasound group — the group will be treated with 1,5 W/cm² 6 minutes in each side of the lumbar spine in 6 points around the lumbar spine
  Other Names: Sonopulse III; Ibramed; 1 MHz and 3 MHz of frequency
  Arms: Pulsed ultrasound group; low level laser therapy group
Other: pulsed ultrasound group — the group will be treated with 1,5 W/cm² 6 minutes in each side of the lumbar spine in 6 points around the lumbar spine
  Other Names: Sonopulse III; Ibramed; 1 MHz and 3 MHz of frequency
  Arms: Continuous ultrasound group; low level laser therapy group
Other: low level laser therapy group — the group will be treated with 3 J 6 minutes in each side of the lumbar spine in 6 points around the lumbar spine
  Other Names: Laserpulse; Ibramed; 904 nm
  Arms: Continuous ultrasound group; Pulsed ultrasound group

SUMMARY:
The objective of this study is evaluate the laser and ultrasound effect on pain and disability in women with non-specific chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* non-specific chronic low back pain
* moderate pain
* eutrophics women

Exclusion Criteria:

* disk herniation
* cardiac diseases
* psychiatrics diseases
* endocrinous diseases
* fractures of the spine
* fractures of lower members
* diabetics
* dental emergency
* local infections
* local non sensibility
* analgesics and anti-inflammatories in use
* neurologic diseases
* pregnancy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-05; Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Pain evaluation | The pain will be evaluate before and after 25 days of the treatment
  The visual analogic scale will be used for evaluate the pain.

SECONDARY OUTCOMES:
Disability evaluation | The disability will be evaluate before and after 25 days of the treatment
  The Roland Morris questionaire will be used to evaluate the disability.

OTHER OUTCOMES:
Multidimensional evaluation of pain | The multidimensional evaluation of pain will be realized before and after 25 days of the treatment
  The McGill questionaire will be used for the evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: ANA PAULA RUBIRA, MASTER, Principal Investigator — SÃO PAULO UNIVERSITY
Locations (1):
- Sâo Lucas College, Porto Velho, Rondônia, Brazil

REFERENCES:
- [Derived] Rubira APFA, Rubira MC, Rubira LA, Comachio J, Magalhaes MO, Marques AP. Comparison of the effects of low-level laser and pulsed and continuous ultrasound on pain and physical disability in chronic non-specific low back pain: a randomized controlled clinical trial. Adv Rheumatol. 2019 Dec 17;59(1):57. doi: 10.1186/s42358-019-0099-z. PMID 31847915
- [Derived] de Resende Guimaraes MFB, Rodrigues CEM, Gomes KWP, Machado CJ, Brenol CV, Krampe SF, de Andrade NPB, Kakehasi AM. High prevalence of obesity in rheumatoid arthritis patients: association with disease activity, hypertension, dyslipidemia and diabetes, a multi-center study. Adv Rheumatol. 2019 Oct 16;59(1):44. doi: 10.1186/s42358-019-0089-1. PMID 31619287